CLINICAL TRIAL: NCT01228409
Title: An Open Label Trial to Show That Subjects With Severe Plaque-Type Psoriasis Receiving Acitretin 25 mg/Day And Stabilized On A Photochemotherapy Regimen Who Are Experiencing Retinoid-Related Adverse Events, Benefit From A Reduction In Acitretin Dose to 17.5 mg/Day, While Maintaining Comparable Efficacy Along With Improved Tolerability
Brief Title: Low-Dose (17.5 mg/Day) Acitretin: Comparable Efficacy Without the Side Effects?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frankel, Amylynne, M.D. (Other)
Collaborators: Stiefel, a GSK Company (Industry)
Responsible Party: Amylynne Frankel, MD, Dermatopharmacology Fellow, Mount Sinai School of Medicine, Department of Dermatology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDAAA 10-0093
Record Dates: First submitted 2010-10-21; First posted 2010-10-26 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Psoriasis
Keywords: Psoriasis; phototherapy; soriatane; acitretin; retinoid-related adverse events
MeSH Terms: conditions — Psoriasis | interventions — Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low dose Acitretin (17.5 mg) (Other)
  Interventions: Drug: Acitretin 17.5 mg/day

INTERVENTIONS:
Drug: Acitretin 17.5 mg/day — lower dose of Acitretin to 17.5 mg/day from 25 mg/day in those experiencing retinoid-related side effects
  Other Names: soriatane, acitretin

SUMMARY:
Psoriasis is a chronic skin disorder with a prevalence of approximately 1-3% worldwide. At present, there is no curative therapy available and the clinical course is unpredictable, but in the majority of cases psoriasis is a chronically remitting and relapsing disease. Several clinical subtypes of psoriasis exist with differences in manifestations and skin areas involved.

Chronic stable plaque psoriasis (Psoriasis Vulgaris) is the commonest form of the disease, accounting for 85-90% of cases. The circumscribed infiltrated skin lesions are scaly and erythematous and often symmetrically distributed over the body. Several types of palliative therapies exist. The therapies are either topical or systemic. The severity of chronic plaque psoriasis is often determined by the percentage of body surface area (BSA) involved. For mild, moderate and severe chronic plaque psoriasis with BSA involvement of up to 20%, initial therapy is topical. Phototherapy and numerous systemic therapies are usually indicated when more than 20% of skin is affected.

Severe plaque-type psoriasis requires systemic and long-term therapy in order to induce and maintain remission. Acitretin 25mg/day combined with a phototherapy regimen is a standard treatment that provides clinically significant efficacy, however many patients experience tolerability issues due to retinoid-related adverse events. Retinoid-related adverse events include but are not limited to: alopecia, dry mucus membranes, pruritus, photosensitivity, elevation of liver enzymes, elevation of serum triglycerides, cholesterol and decrease of HDL, arthralgias, myalgias, eye irritation, blepharitis, photophobia, conjunctivitis, headaches, nausea, anemia and leukemia. Reducing the acitretin dose from 25mg/day to 17.5mg/day may provide improved tolerability without compromising efficacy.

The purpose of this study is to ascertain if reducing the acitretin dose from 25mg/day to 17.5mg/day will provide improved tolerability without compromising efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older.
* Surgically sterile females. Females who have had a hysterectomy or oophorectomy or completed menopause (post-menopausal for at least 1 year) are allowed. Men must agree to use 2 forms of birth control (eg condoms, spermicide).
* Stabilized on a phototherapy regimen for 4 weeks.
* Compliant with acitretin dosing at 25 mg/day and experiencing retinoid-related adverse events which, in the clinical judgement of the investigator, may benefit from a reduction in dose to 17.5 mg/day.
* Able to complete the study and to comply with the study instructions.
* Adherence to alcohol avoidance during acitretin therapy and for 2 months after discontinuation of acitretin.
* Subjects must be willing to not donate blood during the study as well as 3 years following completion of this study.
* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.

Exclusion Criteria:

* Uncontrolled hypertriglyceridemia.
* Guttate, erythrodermic, or pustular psoriasis.
* Severely impaired hepatic function, > 3 times the upper limit of normal and the clinical investigator's judgment.
* Use of systemic immunosuppressant agents (eg. Methotrexate, cyclosporine, thioguanine, azathioprine, alefacept, egalizumab, corticosteroids) within 4 weeks of baseline and throughout the study.
* Topical vitamin A, vitamin D or analogue preparations, or anthralin within 2 weeks of study initiation.
* History of known or suspected intolerance to any of the ingredients of the investigational study product.
* Used over the counter (non-prescription) medications or herbal remedies within 2 weeks of dosing, unless agreed upon as not clinically relevant by the principal investigator.
* Participated in a previous study of the same study product.
* Currently using any medication which, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
* Currently suffering from any disease or condition which, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
* Any major illness within 30 days before screening examination.
* Considered immunocompromised.
* A clinically relevant history of or current evidence of abuse of alcohol or other drugs.
* Use of any investigational drugs or treatments during the study or within 4 weeks of the baseline visit.
* Women of child-bearing potential (see inclusion criteria).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in psoriasis | 12 weeks
  Improvement and maintenance of Psoriasis Area Severity Index (PASI), Body Surface Area (BSA), Physician's Global Assessment (PGA), and Psoriasis Disability Index and Dermatology Life Quality Index (DLQI)

SECONDARY OUTCOMES:
Subjective efficacy/tolerability | 12 weeks
  Subjective efficacy/tolerability questionnaires for every subject at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Clinical Trials, New York, New York, United States